CLINICAL TRIAL: NCT06071520
Title: Andalusian Experience in the Use of Fostamatinib in Patients With ITP. FOSTASUR Study
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FOSTASUR
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — fostamatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PTI patients treated with fostamatinib: Patient with criteria of PTI who has been treated with fostamatinib in the time described
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Patient treated with fostamatinib in the period described
  Other Names: Andalusian PTI fostamatinib patients

SUMMARY:
Description of the use of fostamatinib in patients with PTI in the Andalusian region.

DETAILED DESCRIPTION:
Fostamatinib is a splenic tyrosine kinase (SYK) inhibitor whose indications include the treatment of chronic primary immune thrombocytopenia (PTI) refractory to first-line treatments. Data from two phase 3 studies in PTI, together with supporting safety data from a comprehensive program in 3,437 subjects with rheumatoid arthritis, led to the approval and registration of fostamatinib by health authorities in the US and in Europe.

Given the recent commercialization of fostamatinib for PTI, there is little data in real clinical practice that helps its general management: how to perform tapering, response rates in less refractory patients, experience in subjects with associated immunosuppressive therapies or thrombopoietin analogues, etc. These studies outside the clinical trial environment are relevant to plan needs, consumption, efficacy, and safety results in real clinical practice in our environment, the Andalusian region. The pivotal studies present experience on 102 cases and the real-life experience is of case series of less than 5 patients, with the population of patients treated in the Andalusian region as of December 31st being greater than 40 cases. For all these reasons the Andalusian Group of Congenital Coagulopathies proposes collecting what the experience has been like in their environment. Participation in this study is not intended to change the routine treatment patients receive as determined by their prescribing physicians. No clinic visits, procedures, evaluations, or tests will be required for the purposes of the study. This is multicenter retrospective data that will be collected from information generated during routine examinations and treatments performed by the investigator according to the standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older.
2. Patients with ITP criteria according to clinical practice guidelines.

Exclusion Criteria:

1. Patients with any medical or psychological condition that prevents them from following the procedures of normal clinical practice as determined by the investigator.
2. Subjects with other concomitant hemostatic defects.
3. Documented history or clinical evidence of medical conditions (other than ITP) that consider the underlying cause of thrombocytopenia.
4. Diagnosis of secondary immune thrombocytopenia.
5. Subject has a known allergy to fostamatinib or any of the ingredients included in its formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with fostamatinib for ITP between October 2021 (marketing date in Spain) and December 2022 in the Andalusian region.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Description of fostamatinib use | From fostamatinib prescription first date
  Description of dose and treatment duration of fostamatinib in patients primary immune thrombocytopenia (PTI)

SECONDARY OUTCOMES:
Response | Whenever it occurs after the start of treatment with fostamatinib
  Platelets count greater than 30x10^9/L and greater than 50X10^9/L at least once during treatment in the absence of combination treatment or rescue therapy.
Response duration | Whenever it occurs after the start of treatment with fostamatinib
  Duration in weeks of response greater than 30x10^9/L, 50x10^9/L and 100x10^9/L.
Response failure rate | Whenever it occurs after the start of treatment with fostamatinib
  Platelets count less than 30x10^9/L after four weeks of treatment.
Efficiency | Whenever it occurs after the start of treatment with fostamatinib
  Identify situations that limits the effectiveness of fostamatinib.
Rescue treatment | Whenever it occurs after the start of treatment with fostamatinib
  Percentage of patients who required rescue therapy.
Associated therapies | Whenever it occurs after the start of treatment with fostamatinib
  Percentage of patients who have required therapy for ITP associated with fostamatinib.
Bleeding | Whenever it occurs after the start of treatment with fostamatinib
  Description of hemorrhagic events.
Side effects | Whenever it occurs after the start of treatment with fostamatinib
  Description of side effects associated with the use of fostamatinib.
Security | Whenever it occurs after the start of treatment with fostamatinib
  Number of emergencies, unscheduled visits or hospitalizations for PTI related causes during treatment with fostamatinib.

CONTACTS AND LOCATIONS:
Overall Officials: María Eva Mingot Castellano, MD-PhD, Principal Investigator — Universisty Hospital Virgen del Rocío
Locations (14):
- Spain (14):
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital de Puerto Real, Puerto Real, Cádiz
  - Hospital de Riotinto, Minas de Ríotinto, Huelva
  - Hospital de la Serranía de Ronda, Ronda, Málaga
  - Hospital de la Merced de Osuna, Osuna, Sevilla
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario de Jaén, Jaén
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: Yes
Summaries or oral presentations will be presented with descriptive, preliminary results, by subgroups and finals of the study at international and national congresses of Hematology Societies.